CLINICAL TRIAL: NCT00033410
Title: A Phase I Study Of Tirapazamine (NSC 130181) Paclitaxel And Carboplatin With Concurrent Radiation Followed By Tirapazamine/Paclitaxel/Carboplatin Consolidation For Stage III Non-Small Cell Lung Cancer
Brief Title: Chemotherapy, Tirapazamine, and Radiation Therapy in Treating Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: California Cancer Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069281; CCC-PHI-31; CHNMC-PHI-31; NCI-571
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2006-09

CONDITIONS: Lung Cancer
Keywords: stage II non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Carboplatin; Paclitaxel; Tirapazamine; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel
Drug: tirapazamine
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Tirapazamine may make the tumor cells more sensitive to radiation therapy. Combining chemotherapy, radiation therapy, and tirapazamine may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining chemotherapy with tirapazamine and radiation therapy in treating patients who have stage II or stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of tirapazamine when administered with paclitaxel, carboplatin, and concurrent radiotherapy in patients with stage IIB-IIIB non-small cell lung cancer.
* Determine, preliminarily, the response rate and survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter, dose-escalation study of tirapazamine.

Patients receive induction chemotherapy comprising tirapazamine IV over 2 hours and carboplatin IV over 30 minutes on days 1, 8, 15, 22, 29, and 36 and paclitaxel IV over 1 hour on days 1, 4, 8, 11, 15, 18, 22, 25, 29, 32, 36, and 39. Beginning on day 1, patients undergo radiotherapy once daily 5 days a week for 6.5 weeks. Beginning 4-5 weeks after completion of radiotherapy, patients with stable or responding disease receive consolidation chemotherapy comprising paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on days 1 and 22.

Cohorts of 3-6 patients receive escalating doses of tirapazamine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: Approximately 3-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed primary bronchogenic non-small cell lung cancer

  * Adenocarcinoma
  * Large cell carcinoma
  * Squamous cell carcinoma
* Stage IIIA or IIIB disease (T1-4, N2-3)

  * Mediastinal lymph nodes at least 2 cm in diameter by radiography sufficient to stage N2-3 (must be node positive [cytologically or histologically confirmed] if largest mediastinal node is less than 2 cm in diameter) OR
* Selected stage IIB disease (T3, N0 or T3, N1 with a medical condition that precludes surgery)

  * No malignant pleural effusion
* Measurable or evaluable disease by chest x-ray or CT scan

  * No metastatic disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-2 OR
* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,500/mm^3
* Platelet count normal

Hepatic:

* Not specified

Renal:

* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No uncontrolled congestive heart failure
* No unstable angina
* No unstable cardiac arrhythmias

Pulmonary:

* FEV_1 at least 1.0 L

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No clinically significant hearing loss

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for lung cancer

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for lung cancer

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2002-03

CONTACTS AND LOCATIONS:
Overall Officials: Derick H. Lau, MD, Study Chair — University of California, Davis
Locations (2):
- United States (2):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California Davis Cancer Center, Sacramento, California